CLINICAL TRIAL: NCT05655299
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VTX958 in Participants With Moderate to Severe Psoriasis
Brief Title: VTX958 Versus Placebo for the Treatment of Moderate to Severe Psoriasis
Acronym: Serenity PsO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Ventyx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX958-201
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis
Keywords: TYK2 inhibitor; moderate to severe psoriasis; Ventyx; VTX958
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will employ a double-blind design. Subjects, Investigators, study center staff, persons performing the assessments, and the Sponsor are to remain blinded to the identity of the study treatment from the time of randomization until the database lock for the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VTX958 Dose A (Experimental)
  Interventions: Drug: VTX958 Dose A
- VTX958 Dose B (Experimental)
  Interventions: Drug: VTX958 Dose B
- VTX958 Dose C (Experimental)
  Interventions: Drug: VTX958 Dose C
- VTX958 Dose D (Experimental)
  Interventions: Drug: VTX958 Dose D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VTX958 Dose A — Dose A
  Arms: VTX958 Dose A
Drug: VTX958 Dose B — Dose B
  Arms: VTX958 Dose B
Drug: VTX958 Dose C — Dose C
  Arms: VTX958 Dose C
Drug: VTX958 Dose D — Dose D
  Arms: VTX958 Dose D
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study to understand if taking VTX958 is safe and effective in participants diagnosed with moderate to severe psoriasis (PsO). Approximately 200 patients will take VTX958 Dose A, VTX958 Dose B, VTX958 Dose C, VTX958 Dose D, or placebo.

The study consists of a 30-day Screening Period (to see if a participant qualifies for the study), a 16-week double-blind period (a participant receives active Dose A, Dose B, Dose C, Dose D, or placebo), a 16-week Long Term Extension (LTE) period, a 36-week Open Label Extension (OLE) period and a 4-week Follow-Up Period. The maximal duration of treatment will be approximately 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged 18 years or older.
* History of primarily plaque psoriasis for at least 6 months prior to the screening visit.
* Has had stable psoriasis conditions for at least 3 months before screening.
* Has moderate to severe plaque psoriasis as defined by a PASI score of ≥ 12 and an sPGA score of ≥ 3 at screening and Day 1.
* Has plaque psoriasis covering ≥ 10% of the total BSA at screening and Day 1.
* Deemed by the investigator to be eligible for phototherapy or systemic therapy.
* Females of childbearing potential must agree to use a highly effective contraceptive method from at least 4 weeks prior to Day 1 until at least 4 weeks after the last dose of study product.

Exclusion Criteria:

* Female who is breastfeeding, pregnant, lactating, or who is planning to become pregnant during the study.
* Has evidence of erythrodermic, pustular, predominantly inverse or guttate psoriasis, or drug-induced psoriasis.
* History of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
* Participant is known to have immune deficiency or is immunocompromised.
* Has immune-mediated conditions commonly associated with psoriasis, such as psoriatic arthritis, active uveitis, inflammatory bowel disease, that currently require systemic treatment (including corticosteroids, immunosuppressants, or biologics).

Note: Participants with immune-mediated conditions commonly associated with psoriasis that do not require systemic treatment may be included in the study.

* Has used any topical medication that could affect psoriasis (including corticosteroids, retinoids, vitamin D analogues [such as calcipotriol], Janus kinase [JAK] inhibitors, or tar) within 2 weeks prior to Day 1.
* Has used any systemic treatment that could affect psoriasis (including corticosteroids, oral retinoids, immunosuppressive medication, anakinra, methotrexate, cyclosporine, oral JAK inhibitors, or apremilast) within 4 weeks prior to Day 1.

Note: Intranasal corticosteroids and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are also allowed.

* Participant has received any ultraviolet B (UVB) phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day 1.
* Participant has had psoralen and ultraviolet A (PUVA) treatment within 4 weeks prior to Day 1.
* Participant has received treatment with an investigational or marketed TYK2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Proportion of subjects achieving PASI-75 at Week 16
Adverse Event (AE) / Serious Adverse Event (SAE) Incidence Rate through study completion | Screening through study completion, up to 76 weeks
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
Static Physician's Global Assessment (sPGA) Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Proportion of participants achieving a sPGA score of 0 (clear) or 1 (almost clear) at Week 16
PASI Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Change and percent change from baseline in PASI at Week 16
PASI Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Proportion of participants achieving PASI-90 at Week 16
PASI Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Proportion of participants achieving PASI-100 at Week 16
Dermatology Life Quality Index (DLQI) Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Change from baseline in DLQI scores at Week 16
Body Surface Area (BSA) Efficacy at 16 weeks | Day 1 of Placebo-controlled treatment period to week 16
  Change from baseline in BSA at Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Naik, PhD, Study Director — Ventyx Biosciences, Inc
Locations (63):
- United States (38):
  - Local Site # 840012, Birmingham, Alabama
  - Local Site # 840006, Birmingham, Alabama
  - Local Site # 840028, Phoenix, Arizona
  - Local Site # 840032, Bryant, Arkansas
  - Local Site # 840041, North Little Rock, Arkansas
  - Local Site # 840031, Fountain Valley, California
  - Local Site # 840026, Lomita, California
  - Local Site # 840019, Santa Rosa, California
  - Local Site # 840003, Sherman Oaks, California
  - Local Site # 840040, Boca Raton, Florida
  - Local Site # 840011, Doral, Florida
  - Local Site # 840023, Hialeah, Florida
  - Local Site # 840021, Miami Lakes, Florida
  - Local Site # 840044, North Miami Beach, Florida
  - Local Site # 840010, Ocala, Florida
  - Local Site # 840004, Tampa, Florida
  - Local Site # 840001, Tampa, Florida
  - Local Site # 840045, West Palm Beach, Florida
  - Local Site # 840029, Marietta, Georgia
  - Local Site # 840035, Clarksville, Indiana
  - Local Site # 840005, Indianapolis, Indiana
  - Local Site # 840030, Plainfield, Indiana
  - Local Site # 840013, Louisville, Kentucky
  - Local Site # 840022, Rockville, Maryland
  - Local Site # 840008, Brighton, Massachusetts
  - Local Site # 840016, Bay City, Michigan
  - Local Site # 840007, Fort Gratiot, Michigan
  - Local Site # 840002, Troy, Michigan
  - Local Site # 840034, New Brighton, Minnesota
  - Local Site # 840024, Saint Joseph, Missouri
  - Local Site # 840027, Portsmouth, New Hampshire
  - Local Site # 840042, Wilmington, North Carolina
  - Local Site # 840037, Mason, Ohio
  - Local Site # 840009, Portland, Oregon
  - Local Site # 840038, Rapid City, South Dakota
  - Local Site # 840015, Murfreesboro, Tennessee
  - Local Site # 840039, Pflugerville, Texas
  - Local Site # 840014, Spokane, Washington
- Canada (9):
  - Local Site # 124012, Fredericton
  - Local Site # 124010, Mississauga
  - Local Site # 124002, Montreal
  - Local Site # 124004, North Bay
  - Local Site # 124011, Oshawa
  - Local Site # 124007, Peterborough
  - Local Site # 124008, Québec
  - Local Site # 124005, Toronto
  - Local Site # 124006, Windsor
- Poland (16):
  - Local Site # 616015, Bialystok
  - Local Site # 616016, Bialystok
  - Local Site # 616001, Katowice
  - Local Site # 616014, Krakow
  - Local Site # 616004, Lodz
  - Local Site #616010, Lublin
  - Local Site # 616011, Mikołów
  - Local Site # 616009, Nowa Sól
  - Local Site # 616003, Ostrowiec Świętokrzyski
  - Local Site # 616008, Poznan
  - Local Site # 616007, Szczecin
  - Local Site # 616013, Szczecin
  - Local Site # 616005, Warsaw
  - Local Site # 616002, Wroclaw
  - Local Site # 616006, Wroclaw
  - Local Site # 616018, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided